CLINICAL TRIAL: NCT00313248
Title: Phase 2 Study to Investigate the Efficacy and Safety of ZK-Epothilone (ZK-Epo; ZK 219477) in Patients With Metastatic Breast Cancer
Brief Title: Evaluation of a New Agent for Treatment of Advanced Stage Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 91466; 307975 (Other: company internal)
Record Dates: First submitted 2006-04-11; First posted 2006-04-12 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-11

CONDITIONS: Breast Neoplasm
Keywords: Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — sagopilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Sagopilone (ZK 219477)
- Arm 2 (Experimental)
  Interventions: Drug: Sagopilone (ZK 219477)

INTERVENTIONS:
Drug: Sagopilone (ZK 219477) — All patients will receive ZK-Epo at a dose of 16mg/m2 as an intravenous infusion. Chemotherapy for recurrent breast cancer.
  Other Names: BAY86-5302
  Arms: Arm 1
Drug: Sagopilone (ZK 219477) — Patients will receive 22mg/m2 as intravenous infusion.
  Other Names: BAY86-5302
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate whether treatment with a new drug called ZK-Epothilone (ZK-Epo) in patients with metastatic breast cancer helps to decrease or stop tumor growth.

DETAILED DESCRIPTION:
This study has previously been registered by Berlex, Inc. Berlex, Inc. has been renamed to Bayer HealthCare Pharmaceuticals, Inc.Bayer HealthCare Pharmaceuticals, Inc.is the sponsor of this study.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer (meaning the cancer has spread beyond its original location)
* At least one measurable lesion by CT or MRI
* Progression of disease following previous therapy for breast cancer
* Have received previous treatment with anthracyclines (e.g. doxorubicin[Adriamycin or Doxil] or epirubicin [Ellence]), taxanes (paclitaxel [Taxol or Abraxane] or docetaxel [taxotere]) for your breast cancer
* Not be pregnant
* Additional criteria to be determined at screening visit.

Exclusion Criteria:

* More than 3 previous chemotherapy regimens
* More than one treatment with non cytotoxic agents for breast cancer therapy (e.g. herceptin [trastuzumab] or Avastin [bevacizumab)
* Prior treatment with epothilones (e.g. Ixabepilone)
* Symptomatic brain metastases
* Additional criteria to be determined at screening visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Response to treatment with ZK-Epo after 6 cycles | complete or partial response after 2 to 6 courses of therapy.

SECONDARY OUTCOMES:
Safety and tolerability of ZK-Epo | time to progression after start of study treatment and response duration from time between first date of confirmed PR or CR.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (25):
- United States (21):
  - Birmingham, Alabama
  - Anchorage, Alaska
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Bakersfield, California
  - Palm Springs, California
  - Aurora, Colorado
  - Washington D.C., District of Columbia
  - Daytona Beach, Florida
  - Decatur, Illinois
  - New Albany, Indiana
  - Baltimore, Maryland
  - Minneapolis, Minnesota
  - Livingston, New Jersey
  - New York, New York
  - Syracuse, New York
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Houston, Texas
  - San Antonio, Texas
  - Tacoma, Washington
- Canada (4):
  - Toronto, Ontario
  - Greenfield Park, Quebec
  - Montreal, Quebec
  - Québec, Quebec

REFERENCES:
- [Derived] Morrow PK, Divers S, Provencher L, Luoh SW, Petrella TM, Giurescu M, Schmelter T, Wang Y, Hortobagyi GN, Vahdat LT. Phase II study evaluating the efficacy and safety of sagopilone (ZK-EPO) in patients with metastatic breast cancer that has progressed following chemotherapy. Breast Cancer Res Treat. 2010 Oct;123(3):837-42. doi: 10.1007/s10549-010-1102-x. Epub 2010 Aug 10. PMID 20697802